CLINICAL TRIAL: NCT06200428
Title: The Effect of the Pregnancy Pillow Used in the Last Trimmester on Fatigue and Comfort: Randomized Controlled Study)
Brief Title: The Effect of the Pregnancy Pillow Used in the Last Trimmester on Fatigue and Comfort
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AmasyaU-betuluzun-003
Record Dates: First submitted 2023-12-28; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Sleep Support Pillow
Keywords: Pregnancy; sleep support pillow; sleep; fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): First of all, the pregnant women included in the experimental group;
  * Survey forms and scales will be applied in the pre-test (in weeks 29-30).
  * Then, a pregnancy pillow will be given and necessary explanations will be given about its use.
  * Second follow-up 33-34. It will be done during the first week of pregnancy and the scales will be repeated.
  * The last test is 37-38. It will be done during the gestational week (before birth) and the research will be completed.
  * Pregnancy pillow provides support and relief to 5 different parts of the body simultaneously.
  * It protects the health of expectant mothers during pregnancy and helps reduce neck, abdominal, waist, back and leg pain.
  * It does not lose its shape, become felt or flat with use.
  * Thanks to its zipper, the cover can be easily removed and washed, and can be put on just as easily.
  Interventions: Other: sleep support pillow
- Control group (No Intervention): To the pregnant women included in the control group, the researcher;
  * The survey forms and scales will be applied in the pre-test and no other intervention will be applied (in weeks 29-30).
  * Pregnant women in the control group were given 33-34 and 37-38 days. The last test will be done in a week.

INTERVENTIONS:
Other: sleep support pillow — A sleep support pillow will be used in this study.
  Arms: Experimental group

SUMMARY:
Detecting fatigue experienced during pregnancy and intervening with an effective intervention has an important place in both improving the comfort during pregnancy and the healthy progress of pregnancy, birth and postpartum period. Determining the severity of fatigue experienced during pregnancy and identifying risk factors can help midwives design adequate and effective interventions for pregnant women in this sensitive period (Çoban & Yanıkkerem, 2010; Türkmen, 2014).

The planned research was aimed to examine the effect of the pregnancy pillow used in the last trimester on fatigue and comfort.

DETAILED DESCRIPTION:
Pregnancy is a natural and physiological event. However, the physiological, psychological and metabolic changes that occur in this process may bring about some disorders (Şahin & Kiliçarslan, 2010; Yanikkerem, Altiparmak, & Karadenİz, 2006). Disorders that occur during this period may differ depending on the week of pregnancy. In the first trimester, breast tenderness, nausea-vomiting, frequent urination; in the second trimester; Constipation, headache, increased appetite, back pain and fatigue may occur (Aydın Özkan, Kaya Şenol, & Aslan, 2020). In the third trimester, due to changing anatomical and physiological changes, edema, frequent urination, muscle cramps, lower back pain, insomnia, shortness of breath, weakness and fatigue may be observed (Aydın Özkan et al., 2020). Fatigue is a condition that is frequently seen, especially in the third trimester of pregnancy, and has an impact on the ability to continue activities of daily living. Although the real cause is unknown, fatigue and weakness can occur in any period of pregnancy. It has also been stated in the literature that it may cause labor pain or postpartum depression (Mortazavi & Borzoee, 2019). Therefore, preventing fatigue during pregnancy is very important.

Comfort is the state of being stress-free and comfortable physiologically, spiritually and socially (Kolcaba & Dimarco, 2005). A woman who completes her pregnancy comfortably has a high sense of self-confidence and quality of life. In the opposite case, it is known that stress, anxiety and depression are experienced more and pregnancy and birth complications increase (Nakamura et al., 2015). Therefore, it is important to determine the comfort levels of pregnant women and know the affecting factors (Aydın Özkan et al., 2020).

Midwives have important duties to improve maternal and indirectly public health by reducing pregnancy problems experienced by women. Midwives should not only provide physical care to pregnant women during prenatal care. Midwives must also fulfill their roles and responsibilities of observation, support, assistance, continuing education and consultancy. Midwives should carefully listen to the symptoms and problems stated by the pregnant woman and determine the extent of the problems. One of the most important problems experienced during pregnancy is fatigue (Cheng et al., 2015; Çoban & Yanıkkerem, 2010; Perry et al., 2014). However, unfortunately, there is no systematic intervention to prevent or treat fatigue experienced during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age,
* Volunteer to participate in the research,
* Primiparous,
* 29-30. week of pregnancy,
* Speaks Turkish,
* At least primary school graduate,
* It is planned to include pregnant women who do not have any chronic, visual/mental or diagnosed psychiatric problems and who do not use medication.

Exclusion Criteria:

* Younger than 18,
* Those who do not volunteer to participate in the research,
* Multiparous,
* Less than 29 weeks,
* Those who do not speak Turkish,
* Illiterate,
* It is planned to exclude pregnant women who have any chronic, visual/mental or diagnosed psychiatric problems and who use medication.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-01-22 (Estimated); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Prenatal comfort scale | baseline and 4 weeks
  The comfort is one of the primary outcomes. The comfort levels of pregnant women will be measured using the Prenatal Comfort Scale (PCS).
  The PCS consists of 15 items and 5 sub-dimensions. The scale is evaluated over a total of 75 points. It is interpreted that as the score decreases, the comfort level also decreases, and as the score increases, the comfort level also increases.
Prenatal Comfort Scale (PCS): 2 months | At the end of the 2 months
  From the third trimester, pregnant women will be allowed to sleep on the pregnant pillow. At the end of the 2nd month, PCS will be repeated in order to determine the effect of the pillow used on the sleep and comfort of the pregnant women.
Chalder Fatigue Scale | baseline and 4 weeks
  The scale consists of 11 items in total, including a 7-item physical fatigue subsection and a 4-item mental fatigue subsection. The scale is a four-point Likert type; Less than usual = 0, as much as usual = 1, more than usual = 2, much more than usual = 3. Scoring of the scale can be done in two different ways. Frequently used; It is a scoring between 0-3 and the total score varies between 0-33. This option will be preferred when evaluating the data obtained from the research. In alternative scoring, the first two columns (less than usual, as much as usual) are scored as "0", and the last two columns (more than usual, much more than usual) are scored as "1". High scores indicate greater fatigue severity. When the Cronbach alpha value was examined, it was found that the overall scale had an acceptable level of internal consistency (Cronbach alpha = 0.70).
Chalder Fatigue Scale | At the end of the 2 months
  The scale consists of 11 items in total, including a 7-item physical fatigue subsection and a 4-item mental fatigue subsection. The scale is a four-point Likert type; Less than usual = 0, as much as usual = 1, more than usual = 2, much more than usual = 3. Scoring of the scale can be done in two different ways. Frequently used; It is a scoring between 0-3 and the total score varies between 0-33. This option will be preferred when evaluating the data obtained from the research. In alternative scoring, the first two columns (less than usual, as much as usual) are scored as "0", and the last two columns (more than usual, much more than usual) are scored as "1". High scores indicate greater fatigue severity. When the Cronbach alpha value was examined, it was found that the overall scale had an acceptable level of internal consistency (Cronbach alpha = 0.70).

IPD SHARING:
Plan to Share IPD: No